CLINICAL TRIAL: NCT04557384
Title: A Phase 1, Nonrandomized, Open-Label Investigation of Subcutaneous Ramucirumab Administration in Participants With Advanced Solid Tumors
Brief Title: A Study of Ramucirumab (LY3009806) Given by Injection Under the Skin in Participants With Advanced Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated due to inadequate PK profile associated with the subcutaneous formulation.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17800; I4T-MC-JVDU (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-09-16; First posted 2020-09-21 (Actual); Results first posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Advanced Solid Tumor
Keywords: Safety
MeSH Terms: interventions — Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ramucirumab (Experimental): Participants received starting dose of 700 milligram (mg) ramucirumab loading dose (LD) subcutaneously (SC) followed, a week later, by 350 mg ramucirumab maintenance dose (MD) administered SC once a week.
  Interventions: Drug: Ramucirumab

INTERVENTIONS:
Drug: Ramucirumab — Administered SC
  Other Names: LY3009806

SUMMARY:
The purpose of this study in participants with advanced cancer is to learn more about the safety of ramucirumab when given by injection under the skin (subcutaneous injection). The study will also measure how much ramucirumab gets into the bloodstream and how long it takes the body to get rid of it.

ELIGIBILITY:
Inclusion Criteria:

* Have evaluable disease per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1).
* In the judgment of the investigator, be an appropriate candidate for experimental therapy and:

  * For Cohort A only: Have exhausted all anticancer treatments with proven clinical benefit OR
  * For Cohorts B and C only: Must have one of the three conditions below:

    * Have exhausted all anti-cancer treatments with proven clinical benefit, OR
    * Have hepatocellular carcinoma or gastric cancer who have received prior treatment, and where IV ramucirumab monotherapy is clinically acceptable treatment after progression OR
    * Have a diagnosis for which IV ramucirumab in combination with additional anticancer therapy is clinically acceptable treatment
    * Additionally, it must be clinically acceptable to delay initiation of the combination partner for 3 weeks from the initiation of ramucirumab dosing.
* Eastern Cooperative Oncology Group performance status score of 0 or 1.
* Have discontinued all previous treatments for cancer with adequate wash-out period and recovered from the acute effects of therapy.
* Have adequate hematologic, hepatic, and renal functions and electrolytes.
* Males and females of child-bearing potential must agree to use highly effective contraceptive methods during study treatment and for at least 84 days/12 weeks following the last dose of study drug.

Exclusion Criteria:

* Have uncontrolled hypertension defined as systolic blood pressure (BP) >150 mmHg or diastolic BP >90 mmHg despite standard medical management.
* Have significant bleeding disorders or experienced Grade 3/4 gastrointestinal (GI) bleeding within 3 months prior to enrollment.
* Have hepatic impairment (such as severe liver cirrhosis Child-Pugh B [or worse], cirrhosis with a history of hepatic encephalopathy, clinically meaningful ascites requiring ongoing treatment with diuretics and/or paracentesis, or history of hepatorenal syndrome).
* Have experienced any arterial thromboembolic events (ATEs), including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina, ≤6 months prior to randomization.
* The participant has clinically relevant congestive heart failure (CHF; New York Heart Association [NYHA] Grade ≥2) or symptomatic or poorly controlled cardiac arrhythmia.
* Have symptomatic central nervous system (CNS) metastases. Screening is not required.
* Have history of GI perforation and/or fistula within 6 months prior to enrollment.
* Have an active uncontrolled systemic bacterial, viral, or fungal infection or serious ongoing uncontrolled intercurrent illness.
* Have a serious or non-healing wound, ulcer, or bone fracture within 4 weeks prior to enrollment.
* Have received IV ramucirumab in the past.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- United States (4):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Oncology Hematology West, Omaha, Nebraska
  - Levine Cancer Institute- Carolinas Medical Center, Charlotte, North Carolina
  - Tennessee Oncology PLLC, Nashville, Tennessee
- Kindai University Hospital, Osaka Sayama-shi, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of Ramucirumab (LY3009806) Given by Injection Under the Skin in Participants With Advanced Cancer — https://trials.lillytrialguide.com/en-US/trial/1KS07d3wTANvMFupLlEcxL

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers included participants who had progressive disease, off protocol therapy due to toxicity and having completed the short-term follow-up, death due to any cause.
Period: Overall Study
Arm/Group | Ramucirumab
Started | 3
Received At Least 1 Dose of Study Drug | 3
Completed | 1
Not Completed | 2
Not completed — Study Terminated by Sponsor | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Ramucirumab: Participants received starting dose of 700 mg ramucirumab LD, SC followed, a week later, by 350 mg ramucirumab MD administered SC once a week.
Arm/Group | Ramucirumab
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.67 (5.508)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Time Curve (AUC) of Ramucirumab
Description: PK: AUC of Ramucirumab over the dosing interval was evaluated. Cycle = 21 days.
Time Frame: Cycle (C) 1 Day (D) 1:Predose; C1D2:24 hours (h) postdose;C1D4:48-96 h postdose;C1D8:predose;C1D15:predose;C1D18:48-96 h postdose;C2D1:predose;C2D8:predose;C2D11:48-96h postdose;C3D1:predose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours/milliliter (ng*hr/mL)
Arm/Group | Ramucirumab
Number analyzed (Participants) | 3
nanograms*hours/milliliter (ng*hr/mL) | NA (NA) — Data were too limited (below the limit of quantification in concentration) and AUC summary was not able to be calculated.

2. Primary Outcome: PK: Maximum Concentration (Cmax) of Ramucirumab
Description: PK: Cmax of Ramucirumab was evaluated.
Time Frame: C1D1:Predose; C1D2:24 hours (h) postdose;C1D4:48-96 h postdose;C1D8:predose;C1D15:predose;C1D18:48-96 h postdose;C2D1:predose;C2D8:predose;C2D11:48-96h postdose;C3D1:predose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Ramucirumab
Number analyzed (Participants) | 3
nanograms per milliliter (ng/mL) | NA (NA) — Data were too limited (below the limit of quantification in concentration) and Cmax was not able to be calculated.

3. Primary Outcome: PK: Serum Trough Concentration (Ctrough) of Ramucirumab
Description: Ctrough of Ramucirumab was evaluated.
Time Frame: C1D8: predose; C1D15: predose; C2D1: predose; C2D8: predose; C3D1: predose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (µg/mL)
Arm/Group | Ramucirumab
Number analyzed (Participants) | 3
microgram per milliliter (µg/mL)
  C1D8 | 12.6 (79)
  C1D15: number analyzed (Participants) | 2
  C1D15 | 20.9 (41.6)
  C2D1: number analyzed (Participants) | 1
  C2D1 | NA (NA) — For n = 1, Individual value = 28.4
  C2D8: number analyzed (Participants) | 1
  C2D8 | NA (NA) — For n = 1, Individual value = 38.3
  C3D1: number analyzed (Participants) | 1
  C3D1 | NA (NA) — For n = 1, Individual value = 34.6

4. Secondary Outcome: Percentage of Participants With Anti-Ramucirumab Antibodies
Description: Percentage of participants with positive treatment emergent anti-drug antibodies was summarized by treatment group. A treatment-emergent ADA (TEADA) was defined as: having a negative ADA at baseline and an ADA titer greater than or equal to 1:20 (that is (i.e.), greater than 2-fold from the minimal required dilution of 1:10) any time post baseline (i.e., treatment-induced); or a 4-fold or greater change in ADA titer from baseline for participants that had a detectable ADA titer at baseline (i.e., treatment boosted).
Time Frame: C1D1: predose; C1D15: predose; C2D8: predose; C4D1: predose
Population: Zero participants were analyzed. Data not collected.
Arm/Group | Ramucirumab
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants With Injection Site Reactions (ISRs)
Description: The number of participants with at least one treatment-emergent injection site reaction is presented. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Cycle 1, Cycle 2, Cycle 3: D1, D8, D15, D22: 5-15 min, 60 min post injection; C1D2: 24 hours (h) post injection; C1D4 (± 1 day)
Population: All randomized participants who received at least one dose of study drug and had at least one post dose safety assessment.
Measure: Number; unit: participants
Arm/Group | Ramucirumab
Number analyzed (Participants) | 3
participants | 1

ADVERSE EVENTS:
Time Frame: Up To 40 Days
Description: All randomized participants who received at least 1 dose of study drug.
Arm/Group | Ramucirumab
All-Cause Mortality (participants affected / at risk) | 1/3
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab (N=3)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab (N=3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)
Fatigue (General disorders) | 1 (1)
Generalised oedema (General disorders) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Lipase increased (Investigations) | 1 (3)
Weight decreased (Investigations) | 1 (1)
Weight increased (Investigations) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Confusional state (Psychiatric disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Embolism (Vascular disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated due to low likelihood of achieving a relevant therapeutic exposure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-26): https://cdn.clinicaltrials.gov/large-docs/84/NCT04557384/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/84/NCT04557384/SAP_001.pdf